CLINICAL TRIAL: NCT05230407
Title: Does BMI Influence Pain Follow vNOTE Surgery
Acronym: BMIVNOTES
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Aya Mohr Sasson, Principal Investigator, The University of Texas Health Science Center, Houston
Other Study IDs: BMIVNOTES-UT
Record Dates: First submitted 2021-12-27; First posted 2022-02-08 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Obese; Surgery; Pain, Postoperative
Keywords: Obesity; Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES); Post-operative pain
MeSH Terms: conditions — Obesity; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women after Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES): Study population will include all women after hysterectomy or adnexal surgery by vNOTE technique
  Interventions: Other: Visual analog scale (VAS) assesment of pain

INTERVENTIONS:
Other: Visual analog scale (VAS) assesment of pain — Post operation VAS score will be assessed before discharge from hospital and 24 hours post operation

SUMMARY:
Overweight and obesity are increasing dramatically worldwide and contribute substantially to the burden of morbidity and mortality. Obesity was considered in the past a relative contraindication for abdominal and pelvic laparoscopy surgeries due to the morbidity that is associated with it. Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) is an emerging field in minimally invasive surgery. By incorporating the advantages of endoscopic surgery, the vNOTES approach avoids abdominal wall wounds and trocar-related complications, including reducing post operation pain.

DETAILED DESCRIPTION:
Introduction

Overweight and obesity are increasing dramatically worldwide and contribute substantially to the burden of morbidity and mortality. The clinical guidelines from the National Heart, Lung, and Blood Institute on the identification, evaluation, and treatment of overweight and obesity in adults recommend that clinicians assess waist circumference of their patients. In concordance to the increase in the prevalence of obesity, waist circumference also has shifted, and a rapid increase in abdominal obesity has been demonstrated.

Obesity was considered in the past a relative contraindication for abdominal and pelvic laparoscopy surgeries due to the morbidity that is associated with it. The major challenges include the difficulty with Verres needle placement, hindered manipulation of laparoscopic instruments, and the accumulation of fat in the omentum that often obstructs the operative field. In addition to complicated anesthesia characterizing obese patients due to reduced supine functional residual capacity, lower chest wall compliance, and increase in carbon dioxide production, pneumoperitoneum created during laparoscopic surgeries adds to increased inspiratory resistance that requires higher minute ventilation rates. Post-operative abdominal pain must be well controlled and avoided because it can further restrict ventilation and prevent ambulation.

Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) is an emerging field in minimally invasive surgery. By incorporating the advantages of endoscopic surgery, the vNOTES approach avoids abdominal wall wounds and trocar-related complications, including reducing post operation pain. Surgical outcomes of total laparoscopic hysterectomy (TLH) and vNOTES hysterectomy in obese patients are in favor for the vNOTES approach considering shorter duration of surgery and postoperative hospitalization, and lower pain scores .

To the best of our knowledge no studies have been published regarding the correlation between BMI to the pain experienced by women following vNOTE surgery. Due to the aforementioned, the aim of our study is to learn whether BMI influence pain following vNOTES.

Material and Methods This is a prospective cohort study conducted in a single tertiary medical center. Study population will include all women planned to undergo vNOTE surgery (hysterectomy or adnexal surgery). Women with previous vaginal operations or combined operations for the treatment of prolapse or urinary complains will be excluded from the study. Demographic and clinical characteristics will be collected from women's medical files. Additionally, operative and post-operative data will be collected including: operation duration, estimated blood loss, operation complications (hypotension, bladder gut or vascular perforation), post-operative complications (hemorrhage, endometritis, vascular - thromboembolic event, ileus).

Primary outcome:

Postoperative visual analogue scale (VAS). Evaluation will be performed before discharge or 24th post operation.

Secondary outcomes:

* Operative and post-operative complication rate
* Operative time
* Pill count
* Time until release

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing vNOTES for hysterectomy or adnexal indication Exclusion Criteria.
* Previous vaginal operation
* Combined current vaginal operation (for the treatment of prolapse/ urinary complaints)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women undergoing vNOTES for hysterectomy or adnexal indication
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Postoperative visual analogue scale (VAS) score | 24 hours after surgery
  Score is scaled between 1(no pain at all) to 10(very strong pain)

SECONDARY OUTCOMES:
Use of medication for pain control | 24 hours after surgery
  The type of medication and the number of pills used

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon author request

REFERENCES:
- [Result] Must A, McKeown NM. The Disease Burden Associated with Overweight and Obesity. 2012 Aug 8. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK279095/ PMID 25905320
- [Result] Mokdad AH, Ford ES, Bowman BA, Dietz WH, Vinicor F, Bales VS, Marks JS. Prevalence of obesity, diabetes, and obesity-related health risk factors, 2001. JAMA. 2003 Jan 1;289(1):76-9. doi: 10.1001/jama.289.1.76. PMID 12503980
- [Result] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Result] Le Bras M, Ribou G, Brachet-Liermain M. [Does mefloquine concentrate in the parasited red cell?]. Presse Med. 1989 Mar 4;18(9):492. No abstract available. French. PMID 2522648
- [Result] Lamvu G, Zolnoun D, Boggess J, Steege JF. Obesity: physiologic changes and challenges during laparoscopy. Am J Obstet Gynecol. 2004 Aug;191(2):669-74. doi: 10.1016/j.ajog.2004.05.077. PMID 15343262
- [Result] Jallad K, Walters MD. Natural Orifice Transluminal Endoscopic Surgery (NOTES) in Gynecology. Clin Obstet Gynecol. 2017 Jun;60(2):324-329. doi: 10.1097/GRF.0000000000000280. PMID 28221179
- [Result] Baekelandt J, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BW, Bosteels JJ. Postoperative outcomes and quality of life following hysterectomy by natural orifice transluminal endoscopic surgery (NOTES) compared to laparoscopy in women with a non-prolapsed uterus and benign gynaecological disease: a systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2017 Jan;208:6-15. doi: 10.1016/j.ejogrb.2016.10.044. Epub 2016 Oct 29. PMID 27880893
- [Result] Baekelandt JF, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol B, Bosteels J. Hysterectomy by transvaginal natural orifice transluminal endoscopic surgery versus laparoscopy as a day-care procedure: a randomised controlled trial. BJOG. 2019 Jan;126(1):105-113. doi: 10.1111/1471-0528.15504. PMID 30325565
- [Result] Kaya C, Yildiz S, Alay I, Aslan O, Aydiner IE, Yasar L. The Comparison of Surgical Outcomes following Laparoscopic Hysterectomy and vNOTES Hysterectomy in Obese Patients. J Invest Surg. 2022 Apr;35(4):862-867. doi: 10.1080/08941939.2021.1927262. Epub 2021 May 26. PMID 34036898